CLINICAL TRIAL: NCT00716586
Title: Treatment of Cystoid Macular Edema in Patients With Retinal Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Gerald A. Fishman, Emeritus Professor of Ophthalmology, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0551
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Retinal Degenerations
MeSH Terms: conditions — Retinal Degeneration | interventions — dorzolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trusopt (2% dorzolamide) (Experimental): Intent to treat population. All participants assigned to Trusopt (2% dorzolamide)
  Interventions: Drug: 2% dorzolamide

INTERVENTIONS:
Drug: 2% dorzolamide — Carbonic anhydrase inhibitor, Trusopt (2% dorzolamide)
  Other Names: Trusopt

SUMMARY:
A small percentage of patients with retinal degeneration accumulate fluid in the center of their retina.

Previous studies using an oral form of treatment has been successful in decreasing this fluid which improves vision.

This study will test the use of a topically applied form of this treatment to the eye to reduce the amount of fluid and improve or preserve vision.

DETAILED DESCRIPTION:
Patients with certain retinal degenerations will be asked to take part in a research study about the use of a topically applied eye drop for treating fluid in the central part of the retina (macular edema).

In the current study, investigators propose to use topical Trusopt in a group of patients with retinal degeneration (RD) to determine its effectiveness in reducing the amount of retinal fluid in patients with RD and macular edema. The methods will involve an initial one month treatment with topical Trusopt three times a day in each eye. After a period of one month, patients will return for a follow-up examination. At baseline, they will have had a measurement of their center vision and a measurement of their macular fluid with a photographic-like procedure termed optical coherence tomography (OCT). After the one month period of treatment, they will again have a measurement of their vision and re-evaluation with OCT. An improvement at least of one line (7 letters) or more of vision will be considered as a clinically significant improvement.

ELIGIBILITY:
Inclusion Criteria:

* Presence of cystic macular fluid on OCT testing

Exclusion Criteria:

* Allergic reaction to sulpha containing compounds
* Intolerance to dorzolamide (Trusopt)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2015-08-11 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald A Fishman, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Walia S, Fishman GA, Molday RS, Dyka FM, Kumar NM, Ehlinger MA, Stone EM. Relation of response to treatment with dorzolamide in X-linked retinoschisis to the mechanism of functional loss in retinoschisin. Am J Ophthalmol. 2009 Jan;147(1):111-115.e1. doi: 10.1016/j.ajo.2008.07.041. Epub 2008 Oct 2. PMID 18834580

RESULTS

PARTICIPANT FLOW:
Groups:
- Trusopt (2 % Dorzolamide).: Topical form of carbonic anhydrase inhibitor, Trusopt (2% dorzolamide), 1 drop three times per day.
Period: Overall Study
Arm/Group | Trusopt (2 % Dorzolamide).
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Topical Form of Carbonic Anhydrase Inhibitor.: Participants 18 years or older with cystoid macular edema and retinal degeneration will be treated with Trusopt.
  dorzolamide: 2% dorzolamide- 1 Gtt TID
Arm/Group | Topical Form of Carbonic Anhydrase Inhibitor.
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants] — Participants will initially be seen by Dr. Fishman and have their foveal thickness, macular fluid and vision measured.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 43
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 42 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Improvement in Foveal Thickness (Macular Fluid) as Measured by Optical Coherence Tomography (OCT)
Description: Foveal thickness measured by OCT. A 17% or greater reduction in foveal thickness was considered an improvement. While initially it was our intent to follow participants at 1, 4, and 7 month intervals, these time periods could not be consistently adhered to based on participant non-compliance with appointments. Consequently, additional participants were subsequently seen at baseline to various time points beyond seven months that ranged from 2 months to 36 months at their most recent visit.
Time Frame: Baseline and most recent visit (2 month up to 36 months)
Population: Intent to treat population (all participants assigned to Trusopt (2% dorzolamide).
Measure: Number; unit: participants
Groups:
- Trusopt (2% Dorzolamide): Topical form of carbonic anhydrase inhibitor, Trusopt (2% dorzolamide), 1 drop three times per day
Arm/Group | Trusopt (2% Dorzolamide)
Number analyzed (Participants) | 44
participants | 36

2. Primary Outcome: Number of Participants With Improvement in Macular Fluid as Measured Subjectively by Optical Coherence Tomography (OCT)
Description: Macular fluid measured subjectively by OCT. A 25% or greater reduction of macular fluid was considered an improvement. While initially it was our intent to follow participants at 1, 4, and 7 month intervals, these time periods could not be consistently adhered to based on participant non-compliance with appointments. Consequently, additional participants were subsequently seen at baseline to various time points beyond seven months that ranged from 2 months to 36 months at their most recent visit.
Time Frame: Baseline and most recent visit (2 months up to 36 months)
Population: Intent to treat population (all participants assigned to Trusopt (2% dorzolamide).
Measure: Number; unit: participants
Groups:
- Trusopt (2% Dorzolamide): Topical form of carbonic anhydrase inhibitor, Trusopt (2% dorzolamide ), 1 drop three times per day.
Arm/Group | Trusopt (2% Dorzolamide)
Number analyzed (Participants) | 44
participants | 36

3. Secondary Outcome: Number of Participants With Improvement of Seven Letters or More Read on a Visual Chart
Description: Visual acuity measured in LogMAR units. Reading 7 letters or more on a visual chart, from baseline to most recent visit, was considered an improvement. While initially it was our intent to follow participants at 1, 4, and 7 month intervals, these time periods could not be consistently adhered to based on participant non-compliance. Consequently, additional participants were subsequently seen at baseline to various time points beyond seven months that ranged from 2 months to 36 months at their most recent visit.
Time Frame: Baseline and most recent visit (2 months up to 36 months)
Population: Intent to treat population (all participants assigned to Trusopt (2 % dorzolamide).
Measure: Number; unit: participants
Arm/Group | Trusopt (2% Dorzolamide)
Number analyzed (Participants) | 44
participants | 20

ADVERSE EVENTS:
Time Frame: Adverse event data will be collected during participant study participation, up to 36 months.
Arm/Group | Topical Form of Carbonic Anhydrase Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No